CLINICAL TRIAL: NCT06728358
Title: Single-centre Prospective Study on the Identification of Clinical, Laboratory, Anatomopathological and Molecular Characteristics for the Future Management of Patients With Neoplasms of the Gastro-intestinal Tract
Brief Title: The Future Management of Patients With Neoplasms of the Gastro-intestinal Tract
Acronym: SOCRATE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 6723
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Adenocarcinoma; Cholangiocarcinoma; Colon Cancer
Keywords: Pancreatic cancer; Bile duct cancer; Colon cancer
MeSH Terms: conditions — Cholangiocarcinoma; Colonic Neoplasms; Pancreatic Neoplasms; Bile Duct Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing molecular analysis (Experimental): Patients undergoing molecular analysis
  Interventions: Diagnostic Test: Molecular analyses

INTERVENTIONS:
Diagnostic Test: Molecular analyses — Search for molecular alterations that correlate with patient prognosis

SUMMARY:
The aim of the present study is to research histological and molecular markers in patients with neoplasia of the gastrointestinal tract.

DETAILED DESCRIPTION:
The aim of the present study is to search for histological and molecular markers in patients with neoplasia of the gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* PS ECOG 0-2;
* Histological diagnosis of cancer of the gastro-enteric district: intestinal, pancreatic, biliary tract neoplasms;
* Radiological evidence of resectable/locally advanced/metastatic disease on the date of the first visit;
* Availability of tumour histological material;
* At least one visit following the first oncological visit.

Exclusion Criteria:

* Absence of histological diagnosis of neoplasm of the gastro-enteric tract;
* Lack of histological specimens on which to perform examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 48 months
  The primary objective of the study is to evaluate the probabilitỳ of survival in terms of OS in relation to the expression of specific anatomopathological, immunohistochemical and molecular markers (GATA6, GemPred Molecular Signature and FOLFIRINOX Molecular Signature) present in the tumour tissue of patients with neoplasms of the gastro-enteric district in the setting of resectable/metastatic disease.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Salvatore, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Policlinico Universitario Agostino Gemelli, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No